CLINICAL TRIAL: NCT00058422
Title: A Phase II Study of R-CHOP and Ibritumomab Tiuxetan (Zevalin) for Elderly Patients With Previously Untreated Diffuse Large B-Cell Lymphoma
Brief Title: Rituximab and Combination Chemotherapy Combined With Yttrium Y 90 Ibritumomab Tiuxetan in Treating Older Patients With Previously Untreated B-Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02-090; MSKCC-02090
Record Dates: First submitted 2003-04-07; First posted 2003-04-09 (Estimated); Results first posted 2020-11-12 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-10

CONDITIONS: Lymphoma
Keywords: noncontiguous stage II adult diffuse large cell lymphoma; stage III adult diffuse large cell lymphoma; stage IV adult diffuse large cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Large B-Cell, Diffuse | interventions — Darbepoetin alfa; Filgrastim; Rituximab; Cyclophosphamide; Doxorubicin; Prednisone; Vincristine; Indium; ibritumomab tiuxetan

ARMS (1):
- R-CHOP and Ibritumomab Tiuxetan (Zevalin) (Experimental): Chemotherapy: Patients receive rituximab IV over 2-5 hours, cyclophosphamide IV, doxorubicin IV, and vincristine IV on day 1; oral prednisone on days 1-5 or 2-6; and filgrastim (G-CSF) subcutaneously (SC) on days 7-15. Patients also receive darbepoetin alfa SC on day 1. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Radioimmunotherapy: Patients receive rituximab IV over 3-5 hours and indium In 111 ibritumomab tiuxetan (IDEC-In2B8) IV over 10 minutes on day 0.
  Patients undergo gamma camera imaging at 2-24 hours and 48-72 hours after the injection of IDEC-In2B8 to observe the flow of ibritumomab tiuxetan. If the flow is deemed safe, then patients receive yttrium Y 90 ibritumomab tiuxetan IV over 10 minutes on day 7. Quality of life is assessed at baseline, before course 5 of chemotherapy, before radioimmunotherapy, and at 3 months. Patients are followed every 3 months for 1 year and then every 6 months for 4 years.
  Interventions: Biological: darbepoetin alfa; Biological: filgrastim; Biological: rituximab; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: prednisone; Drug: vincristine sulfate; Radiation: indium In 111 ibritumomab tiuxetan; Radiation: yttrium Y 90 ibritumomab tiuxetan

INTERVENTIONS:
Biological: darbepoetin alfa
Biological: filgrastim
Biological: rituximab
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: prednisone
Drug: vincristine sulfate
Radiation: indium In 111 ibritumomab tiuxetan
Radiation: yttrium Y 90 ibritumomab tiuxetan

SUMMARY:
RATIONALE: Monoclonal antibodies such as rituximab and yttrium Y 90 ibritumomab tiuxetan can locate cancer cells and either kill them or deliver radioactive cancer-killing substances to them without harming normal cells. Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining rituximab and combination chemotherapy with yttrium Y 90 ibritumomab tiuxetan may kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of combining rituximab and combination chemotherapy with yttrium Y 90 ibritumomab tiuxetan in treating older patients who have B-cell lymphoma that has not been previously treated.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the progression-free and overall survival of patients age 60 and over with previously untreated diffuse large B-cell lymphoma treated with rituximab, cyclophosphamide, doxorubicin, vincristine, and prednisone (R-CHOP) combined with yttrium Y 90 ibritumomab tiuxetan.
* Determine the incidence of adverse experiences, hematologic toxicity (WBC, hemoglobin, and platelet nadirs; and transfusion requirements), cardiac toxicity (incidence of left ventricular dysfunction and cardiomyopathy by echocardiography), and the development of human antimouse antibody/human anti-chimeric antibody in patients treated with this regimen.
* Determine the predictive value of detecting minimal residual disease by molecular techniques for future relapse/recurrence in patients treated with this regimen.
* Determine the response rate of patients treated with this regimen.
* Determine the red blood cell transfusion requirements, change in hemoglobin from baseline, and incidence of anemia with prophylactic darbepoetin alfa support in patients treated with this regimen.
* Determine the conversion rate to complete remission in patients treated with ibritumomab tiuxetan who achieve a partial remission post-R-CHOP.
* Determine the effect of darbepoetin alfa on the quality of life of these patients.

OUTLINE: This is an open-label, nonrandomized study.

* Chemotherapy: Patients receive rituximab IV over 2-5 hours, cyclophosphamide IV, doxorubicin IV, and vincristine IV on day 1; oral prednisone on days 1-5 or 2-6; and filgrastim (G-CSF) subcutaneously (SC) on days 7-15. Patients also receive darbepoetin alfa SC on day 1. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
* Radioimmunotherapy: Patients receive rituximab IV over 3-5 hours and indium In 111 ibritumomab tiuxetan (IDEC-In2B8) IV over 10 minutes on day 0.

Patients undergo gamma camera imaging at 2-24 hours and 48-72 hours after the injection of IDEC-In2B8 to observe the flow of ibritumomab tiuxetan. If the flow is deemed safe, then patients receive yttrium Y 90 ibritumomab tiuxetan IV over 10 minutes on day 7.

Quality of life is assessed at baseline, before course 5 of chemotherapy, before radioimmunotherapy, and at 3 months.

Patients are followed every 3 months for 1 year and then every 6 months for 4 years.

PROJECTED ACCRUAL: A total of 65 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed diffuse large B-cell lymphoma, including any of the following subtypes:

  * Centroblastic
  * Immunoblastic
  * T-cell/histiocyte-rich
  * Lymphomatoid granulomatosis type
  * Anaplastic large B-cell
  * Plasmablastic
  * Mediastinal
  * Intravascular large B-cell lymphoma
* Previously untreated
* High-intermediate or high-risk disease, defined by an age-adjusted international prognostic index score of 2 or 3 (with 1 point each assigned for a ECOG greater than 1/Karnofsky less than 80%, lactate dehydrogenase greater than normal, and stage III or IV)
* Lymphomas with discordant histology and a diffuse large B-cell component are eligible
* Must have an initial diagnostic specimen that is CD20+
* At least Ann Arbor stage II disease

  * No confinement of disease to an involved-field radiotherapy port (stage I or limited stage II disease)
* Bidimensionally measurable disease with at least 1 lymph node at least 2.0 cm by 2.0 cm by physical examination, CT scan, or positron-emission tomography
* Bone marrow cellularity greater than 15%
* No known brain or leptomeningeal metastases
* No primary effusion lymphomas

PATIENT CHARACTERISTICS:

Age

* 60 and over* NOTE: *Patients 60 to 65 years of age must be deemed ineligible for autologous stem cell transplantation

Performance status

* Karnofsky 50-100%

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Bilirubin no greater than 2.0 mg/dL (except for Gilbert's disease)

Renal

* Creatinine no greater than 1.5 mg/dL* OR
* Creatinine clearance greater than 50 mL/min* NOTE: *Patients not meeting either criterion but who have renal insufficiency directly related to lymphomatous involvement of the kidneys or renal collecting system are allowed

Cardiovascular

* Cardiac ejection fraction at least 50% by echocardiogram
* No acute myocardial infarction within the past 3 months
* No uncontrolled hypertension
* No New York Heart Association class III or IV congestive heart failure
* No unstable angina pectoris

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* HIV negative
* B12 and folate greater than the lower limit of normal
* Transferrin saturation at least 15%
* Ferritin greater than 10 µg/L
* At least 6 weeks since prior RBC donation
* No active seizure disorder

  * Prior seizure disorder allowed if free of antiseizure medication and evidence of seizure activity for the past 5 years
* No concurrent uncontrolled medical problems that would preclude administration of chemotherapy or radioimmunotherapy
* No other concurrent malignancy treated with chemotherapy or radiotherapy except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy

* At least 4 weeks since prior RBC transfusion
* No prior biologic therapy
* No other concurrent biologic therapy

Chemotherapy

* No prior chemotherapy (one course of R-CHOP allowed)
* No other concurrent standard or investigational chemotherapy

Endocrine therapy

* No more than 7 consecutive days of prior steroids (premedication allowed for prior intravenous contrast allergy)
* No other concurrent corticosteroids

Radiotherapy

* No prior radiotherapy

Surgery

* Not specified

Ages: 60 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2003-02-10 (Actual); Primary Completion 2019-11-14 (Actual); Study Completion 2019-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul A. Hamlin, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | R-CHOP and Ibritumomab Tiuxetan (Zevalin)
Started | 65
Completed | 63
Not Completed | 2
Not completed — Not treated | 2

BASELINE CHARACTERISTICS:
Arm/Group | R-CHOP and Ibritumomab Tiuxetan (Zevalin)
Number analyzed (Participants) | 65
Age, Continuous [Median (Full Range); unit: years] | 75 [62 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 62
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 4
  White | 57
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 65

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | R-CHOP and Ibritumomab Tiuxetan (Zevalin)
Number analyzed (Participants) | 65
Participants
  Dead | 32
  Alive | 33

2. Primary Outcome: Progression-free Survival
Time Frame: 2 years
Population: Data were not collected
Arm/Group | R-CHOP and Ibritumomab Tiuxetan (Zevalin)
Number analyzed (Participants) | 0

3. Primary Outcome: Event-free Survival
Time Frame: 2 years
Population: Data were not collected
Arm/Group | R-CHOP and Ibritumomab Tiuxetan (Zevalin)
Number analyzed (Participants) | 0

4. Primary Outcome: Incidence of Adverse Experiences
Description: Determine the incidence of adverse experiences, hematologic toxicity (WBC, hemoglobin, and platelet nadirs; and transfusion requirements), cardiac toxicity (incidence of left ventricular dysfunction and cardiomyopathy by echocardiography), and the development of human antimouse antibody/human anti-chimeric antibody in patients treated with this regimen.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | R-CHOP and Ibritumomab Tiuxetan (Zevalin)
Number analyzed (Participants) | 65
Participants | 65

5. Secondary Outcome: Conversion Rate to Complete Remission
Time Frame: 2 years
Population: Data were not collected
Arm/Group | R-CHOP and Ibritumomab Tiuxetan (Zevalin)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | R-CHOP and Ibritumomab Tiuxetan (Zevalin)
All-Cause Mortality (participants affected / at risk) | 32/65
Serious Adverse Events (participants affected / at risk) | 34/65
Other Adverse Events (participants affected / at risk) | 41/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | R-CHOP and Ibritumomab Tiuxetan (Zevalin) (N=65)
Abdominal pain/cramping (Gastrointestinal disorders) | 1
Cardiac left vent (Cardiac disorders) | 4
Cardiovascular, Arrhythmia other (Cardiac disorders) | 2
Cardiovascular, other (Cardiac disorders) | 2
Colititis (Gastrointestinal disorders) | 4
Dehydration (Metabolism and nutrition disorders) | 1
Delusions (Psychiatric disorders) | 1
Derm, skin other (Skin and subcutaneous tissue disorders) | 3
Diarrhea (Pts w/out col) (Gastrointestinal disorders) | 1
Dizziness (Nervous system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 9
Fever (General disorders) | 1
GI, other (Gastrointestinal disorders) | 1
Hemoglobin (Hgb) (Investigations) | 3
Hypernatremia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Hypotension (Vascular disorders) | 2
Infection w.out neutropenia (Infections and infestations) | 13
Infection with grade 3/4 neut (Infections and infestations) | 3
Infection/Feb Neut-Other (Infections and infestations) | 1
Nausea (Gastrointestinal disorders) | 3
Neurology, other (Nervous system disorders) | 1
Platelets (Investigations) | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3
Pulmonary, other (Respiratory, thoracic and mediastinal disorders) | 1
Supravent arrhythmia (Cardiac disorders) | 2
Thrombosis (Vascular disorders) | 6
Vomiting (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | R-CHOP and Ibritumomab Tiuxetan (Zevalin) (N=65)
Febrile neutropenia (Blood and lymphatic system disorders) | 6
Infection w.out neutropenia (Infections and infestations) | 5
Dehydration (Metabolism and nutrition disorders) | 3
Supravent arrhythmia (Cardiac disorders) | 3
Hemoglobin (Hgb) (Blood and lymphatic system disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 2
Infection with grade 3/4 neut (Infections and infestations) | 2
Nausea (Gastrointestinal disorders) | 2
Platelets (Investigations) | 2
Thrombosis (Vascular disorders) | 2
Cardiovascular, Arrhythmia other (Cardiac disorders) | 1
Colititis (Gastrointestinal disorders) | 1
Diarrhea (Pts w/out col) (Gastrointestinal disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Hypotension (Vascular disorders) | 1
Infection/Feb Neut-Other (Infections and infestations) | 1
Lymphopenia (Investigations) | 1
Pulmonary, other (Respiratory, thoracic and mediastinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2007-09-11): https://cdn.clinicaltrials.gov/large-docs/22/NCT00058422/Prot_SAP_000.pdf